CLINICAL TRIAL: NCT04417933
Title: A Prospective, Single-center, Single-arm, Exploratory Study on the Treatment of Recurrent Glioblastoma With Tumor Electric Fields Treatment System
Brief Title: Tumor Electric Fields Treatment System for Glioblastoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Hunan An Tai Kang Cheng Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202001012
Record Dates: First submitted 2020-05-31; First posted 2020-06-05 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Glioblastoma
Keywords: glioblastoma; tumor electric fields treatment
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor Electric Fields Treatment System (Experimental): Patients have a histologically confirmed diagnosis of supratentorial glioblastoma that is recurrent. All patients will receive Tumor Electric Fields Treatment System.
  Interventions: Device: Tumor Electric Fields Treatment System

INTERVENTIONS:
Device: Tumor Electric Fields Treatment System — Patients wear two pairs of electrodes on the head for 19-22 hours a day. Each patient is required to wear the device as long as possible and not less than 6 months. The treatment has a two-day break for every four weeks.
  Other Names: ASCLU-300

SUMMARY:
This early phase I trial will investigate the safety and feasibility of applying the Tumor Electric Fields Treatment System to subjects with recurrent glioblastoma.

DETAILED DESCRIPTION:
Subjects who have previously completed radiotherapy and at least two cycles of chemotherapy with imaging or pathological evidence of tumor recurrence will receive Tumor Electric Fields Treatment System. The main objective is to evaluate the safety of applying the Tumor Electric Fields Treatment System to subjects with recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of glioblastoma at first surgery (WHO Grade IV, supratentorial location);
* Age between 18 and 65 years, male or female;
* Previously completed radiotherapy and at least two cycles of chemotherapy;
* With imaging or pathological evidence of tumor recurrence;
* Karnofsky performance score (KPS) score ≥ 70 before intervention;
* With a life expectancy more than 3 months;
* Adopted effective contraceptive measures at child-bearing age;
* Provided written informed consent.

Exclusion Criteria:

* Patients unwilling to use the equipment ≥ 18h per day;
* With poor compliance or live too far from the research center, who cannot keep regular follow-up or adjust the electrode position of the treatment equipment, and who refuse to receive follow-up to terminal survival;
* With poor healing of scalp wound, poor scalp condition, large skull defect or other cases where electrodes are not suitable for wearing;
* Within 3 months from radiotherapy;
* Within 4 weeks from the last cycle of chemotherapy;
* Within 4 weeks from surgery for recurrence;
* Participated in other clinical trials.
* Pregnant;
* Epilepsy symptoms not effectively controlled;
* Blood and biochemical indicators in the following range: A. Liver function impairment: AST or ALT > 3 times the upper limit of normal; B. Total bilirubin> upper limit of normal value; C. Renal impairment: serum creatinine>1.7mg /dL (>150 mol/L); D. Coagulopathy: PT or APTT >1.5 times normal; E. Platelets counts < 100x10^9/L; F. Absolute neutrophils count < 1x10^9/L; G. Hemoglobin < 100g/L;
* With severe infectious diseases, such as acute severe infection and HIV positive;
* Other conditions, such as an implanted cardiac pacemaker or deep brain stimulator, severe intracranial edema, increased intracranial pressure resulting in midline shift>5mm, clinically significant papilledema, or reduced level of consciousness, allergy to conductive coupling agent, gel, and other serious life-threatening diseases.
* Other circumstances considered inappropriate to participate in the research by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The treatment-related adverse events | 12 months
  Number of patients who experienced a treatment-related adverse event.
Time to Progression | 12 months
  Time to progression of patients with recurrent glioblastoma.
Overall Survival Rate | 12 months
  Number of patients alive at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China